CLINICAL TRIAL: NCT02249338
Title: Effect of 14-Day Treatment With BIIL 284 BS on Patients With COPD (Double-Blind, Placebo-Controlled, Randomised, Parallel Group Study)
Brief Title: Effect of BIIL 284 BS on Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.10
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — amelubant

ARMS (2):
- BIIL 284 BS (Experimental)
  Interventions: Drug: BIIL 284 BS
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS
  Arms: BIIL 284 BS
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate the effect of 14-day treatment with BIIL 284 BS on sputum neutrophils and specific inflammatory markers in patients with clinically well-defined moderate chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD as defined by the American Thoracic Society criteria. Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 ≤ 70 % of predicted value and FEV1/FVC ≤ 70 % at Screening Visit 1
* Ability to produce an adequate induced sputum sample ad defined by: volume > 1 ml: squamous cells less than 80% and the ability to tolerate the procedure for at least four minutes with no bronchoconstriction ( a fall in FEV1 ≥ 20%)
* Greater than 50% of neutrophils in induced-sputum cells at visit 1. This requirement refers to the neutrophils percentage excluding squamous cells
* Males or females aged 40 to 80 years inclusive.
* Female patients of childbearing potential cannot participate in this study. Female patients participating in this study must meet at least one of the following criteria:

  * surgically sterilized by hysterectomy or bilateral tubal ligation
  * post-menopausal for at least two years
* A smoking history of more than ten pack years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
* Patients must be able to perform pulmonary function tests and maintain records during the study period as required in the protocol
* All patients must sign an Informed Consent Form prior tho participation in the trial, i.e., prior to pre-study washout of their usual pulmonary medications

Exclusion Criteria:

* Culture-documented and/or radiographic evidence and/or antibiotic treatment of an upper or lower respiratory tract infection within the previous 4 weeks or during the baseline period of this study
* Significant diseases other than COPD will be exclude. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study. Patients with inflammatory diseases e.g. rheumatoid arthritis, and those with autoimmune diseases will be excluded
* Clinically significant abnormal baseline haematology, liver function, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded. Laboratory parameters listed in the protocol must be within normal range, or if not, be documented by the investigator as not clinically relevant. The following tests may be outside the normal range to the extent indicated:

  * Aspartate transaminase, Alanine transaminase, Total Bilirubin, Alkaline Phosphatase: 10% > upper limit of normal (ULN)
  * White blood cell count < 3.80 x 10**9/L, Neutrophils < 2.00 x 10**9/L, Platelets < 100 x 10**9/L, Hemoglobin < 12 x g/dL
  * Urea Nitrogen, Creatinine: 10% > ULN
* A recent history (i.e. within six months) of myocardial infarction
* A recent history (i.e. within three months) of refractory heart failure or unstable arrhythmias requiring treatment
* Patients with known active tuberculosis
* A history of cancer within the last five years. Patients with treated basal cell carcinoma or cutaneous squamous cell carcinoma are allowed
* A history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Previous thoracotomy with pulmonary resection. Patients with a history of a thoracotomy without pulmonary resection should be evaluated as per exclusion criterion no. 2
* The use of oral corticosteroids within 4 weeks, or theophyllines and oral or long-acting inhaled beta2-agonists within 2 weeks of visit 1
* A change in pulmonary therapy within the 6 weeks prior to the screening visit 1 in order to control the patient's COPD
* A history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥ 600/mm**3
* A history of and/or current alcohol abuse and/or drug abuse
* Use of an investigational drug within one month or six half-lives (which ever is greater) of the screening visit 1

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1999-10; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Percentage of neutrophils in the induced sputum differential cell count | Baseline, day 14

SECONDARY OUTCOMES:
Percentage of neutrophils in the spontaneous sputum differential cell count | Baseline, day 14
Percentage of neutrophils in the induced sputum differential cell count | Baseline, day 28
Percentage of neutrophils in the spontaneous sputum differential cell count | Baseline, day 28
Differential cell count in induced sputum | Baseline, day 14 and 28
  macrophages, lymphocytes, eosinophils, basophils and epithelial cells
Differential cell count in spontaneous sputum | Baseline, day 14 and 28
  macrophages, lymphocytes, eosinophils, basophils and epithelial cells
Wet weight of spontaneous sputum | Day -6, 0, 6, 13 and 27
  collected over a 24 hours period the day before each clinic visit
Concentration of myeloperoxidase (MPO) in induced sputum | Baseline, day 14 and 28
Concentration of myeloperoxidase (MPO) in spontaneous sputum | Baseline, day 14 and 28
Concentration of neutrophil elastase (NE) in induced sputum | Baseline, day 14 and 28
Concentration of neutrophil elastase (NE) in spontaneous sputum | Baseline, day 14 and 28
Concentration of interleukin-8 (IL-8) in induced sputum | Baseline, day 14 and 28
Concentration of interleukin-8 (IL-8) in spontaneous sputum | Baseline, day 14 and 28
Concentration of leukotriene B4 (LTB4) in induced sputum | Baseline, day 14 and 28
Concentration of leukotriene B4 (LTB4) in spontaneous sputum | Baseline, day 14 and 28
Concentration of albumin in induced sputum | Baseline, day 14 and 28
Concentration of albumin in spontaneous sputum | Baseline, day 14 and 28
Sputum bacterial load of induced sputum | Baseline, day 14 and 28
Sputum bacterial load of spontaneous sputum | Baseline, day 14 and 28
Sputum chemotactic activity of induced sputum | Baseline, day 14 and 28
Sputum chemotactic activity of spontaneous sputum | Baseline, day 14 and 28
Inhibition of blood neutrophil Mac-1 expression | Day 1 and 14
  both unstimulated and LTB4-stimulated
Inhibition of blood neutrophil chemotaxis response to LTB4 | Day 1 and 14
Forced expiratory volume in one second (FEV1) | Pre-treatment on Day 1, pre- and 30 min post-treatment on day 7 and 14
Forced vital capacity (FVC) | Pre-treatment on Day 1, pre- and 30 min post-treatment on day 7 and 14
Forced expiratory flow (FEF25-75%) | Pre-treatment on Day 1, pre- and 30 min post-treatment on day 7 and 14
Peak expiratory flow rate (PEFR) | Pre-treatment on Day 1, pre- and 30 min post-treatment on day 7 and 14
Inspiratory capacity (IC) | Pre-treatment on Day 1, pre- and 30 min post-treatment on day 7 and 14
Slow vital capacity (SVC) | Pre-treatment on Day 1, pre- and 30 min post-treatment on day 7 and 14
Changes in COPD symptom score | Baseline, Day 1, 7 and 14
  dyspnoea, fatigue, orthopnea, paroxysmal nocturnal dyspnoea and cough
Physician's global evaluation of symptoms assessed on a 4-point scale | Baseline, Day 14
Number of patients with adverse events | up to 6 weeks
Plasma concentrations of the analytes | 30 min before, 90 and 240 min after drug administration on day 1 and 14